CLINICAL TRIAL: NCT01562574
Title: A Randomised, Double-blind, Parallel Group, Placebo-controlled Comparison of Recombi-nant Factor VIIa (rFVIIa/ NovoSeven®) With Standard Haemostatic Replacement Therapy, and Standard Haemostatic Replacement Ther-apy Following Cardiac Bypass Surgery for Paediatric Congenital Heart Disease
Brief Title: Activated Recombinant Human Factor VII Following Cardiac Bypass Surgery for Paediatric Congenital Heart Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F7CPB-3343
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Acquired Bleeding Disorder; Cardiac Surgery Requiring Cardiopulmonary Bypass

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Activated recombinant human factor VII (Experimental)
  Interventions: Drug: activated recombinant human factor VII
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: activated recombinant human factor VII — Up to three doses administered after surgery. If bleeding persisted after the third dose of trial product, conventional transfusion would be administered
  Arms: Activated recombinant human factor VII
Drug: placebo — Up to three doses administered after surgery. If bleeding persisted after the third dose of trial product, conventional transfusion would be administered
  Arms: Placebo

SUMMARY:
This trial is conducted in Oceania. The aim of this trial is to investigate the efficacy of activated recombinant human factor VII and standard treatment compared with standard haemostatic replacement therapy in cardiopulmonary bypass (CPB) surgery for paediatric congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained from parent or legal guardian before any trial-related activities. Trial-related activities are any procedure that would not have been performed during normal management of the subject
* Children with complex congenital heart disease requiring corrective surgery with cardiopulmonary bypass (CPB)

Exclusion Criteria:

* Congenital heart disease that does not require CPB surgery

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2002-01; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Time from reversal of heparin with protamine sulphate to chest closure

SECONDARY OUTCOMES:
Number of units/volume of fresh frozen plasma (FFP) and/or platelets and/or red-cell concentrates transfused during surgery and in the post-surgery period
Blood loss
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Parkville, Australia

REFERENCES:
- [Result] Ekert H, Brizard C, Eyers R, Cochrane A, Henning R. Elective administration in infants of low-dose recombinant activated factor VII (rFVIIa) in cardiopulmonary bypass surgery for congenital heart disease does not shorten time to chest closure or reduce blood loss and need for transfusions: a randomized, double-blind, parallel group, placebo-controlled study of rFVIIa and standard haemostatic replacement therapy versus standard haemostatic replacement therapy. Blood Coagul Fibrinolysis. 2006 Jul;17(5):389-95. doi: 10.1097/01.mbc.0000233369.03358.c1. PMID 16788315
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com